CLINICAL TRIAL: NCT05033717
Title: Effects of Tissue Flossing Technique Versus Static Stretching Exercises of Bicep Muscle on Pain, Range of Motion and Function in Athletes With Bicipital Tendinitis
Brief Title: Effects of Tissue Flossing Technique for Bicipital Tendinitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC//0413 Aroofa
Record Dates: First submitted 2021-08-27; First posted 2021-09-05 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Bicipital Tendinitis
Keywords: Flossing; Flexibility; ROM; Prevention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Tissue Flossing Technique
  Interventions: Other: Tissue Flossing Technique
- Group B (Active Comparator): Static Stretching exercises
  Interventions: Other: Static Stretching Technique

INTERVENTIONS:
Other: Tissue Flossing Technique — Subjects will receive tissue-flossing intervention on bicep muscle for 30 sec to 2 min with an occlusion pressure of 100 mmHg.
  After removal of flossing, participants will perform bicep strengthening exercises at an intensity of 30% of 1 RM with 6-8 rep, 4 sets for a single day and 3 days per week for 2 weeks in total.
  Arms: Group A
Other: Static Stretching Technique — Subjects will perform passive static stretching exercises of bicep muscle. Each stretch will last for 30 sec at 100% of stretch intensity with 4 reps for each, 1 set per day and 3 days per week for total duration of two weeks.
  After the application of static stretch, participants will perform bicep strengthening exercises at an intensity of 30% of 1 RM with 6-8 reps, 4 sets for a single day and 3 days per week for 2 weeks in total.
  Arms: Group B

SUMMARY:
This project will be a Randomized control trial conducted to check the effects of tissue flossing technique versus static stretching exercises of bicep muscle on pain, range of motion and function in patients with bicipital tendinitis, so that we can have best treatment option for them. Duration will be of 6 months. Purposive sampling will be done. Subjects fulfilling eligibility criteria from Allied hospital Faisalabad, will be randomly allocated in two groups via lottery method. Baseline assessment will be done. Group A participants will be given baseline treatment along with tissue flossing. Group B participants will be given stretching exercises along with baseline treatment for two weeks, 3 sessions per week. Post intervention assessment will be done via, Numeric pain rating scale(NPRS),Shoulder Pain And Disability Index (SPADI) and goniometric measurements of shoulder ranges. Data will be analyzed by using SPSS version 20.

DETAILED DESCRIPTION:
Inflammation of the bicep tendon is also known as "Bicipital Tendinitis" occurs most commonly in overhead athletes like racquet players, swimmers, gymnasts, tennis players, baseball pitchers, and rowing athletes. Tissue Flossing is a relatively novel practice that initially got recognition in weightlifting athletes. This technique has Japanese origin also known as the "Katsu Technique" or "Blood Flow Restriction technique" BFR. It works on the principle of optimizing the blood circulation to the muscles for fitness, early rehabilitation, and recovery within safe ranges.

The purpose of the current study is to determine the effects of the tissue flossing technique on the physical rehabilitation of bicipital tendinitis. It is a randomized controlled trial with the subjects having a history of bicipital tendinitis, shoulder pain, and recreational athletes with difficulty in overhead activities. Subjects with a history of neurological and psychological disorders, hypertension or heart diseases and with chronic arthritis will be excluded.

Participants will be randomly placed into experimental and control groups. The experimental group will receive bicep-strengthening exercises after flossing. The Control group will receive bicep-strengthening exercises after bicep-stretching exercises. The total duration of this study will be six months with an assessment performed at baseline, before and after the treatment sessions. Numeric Pain rating scale, Goniometer, and Shoulder Pain and Disability Index will be used to measure the outcomes. Data will be analyzed statistically by using parametric or non-parametric tests after the completion of this study.

ELIGIBILITY:
Inclusion Criteria:

* Bicep tendinitis with age 18 to 45 years
* Subjects with a history of repetitive overhead activities and pain in bicipital groove.
* Recent history of adhesive capsulitis.
* Chronic bicep weakness with history of recreational activities.
* Recreational athletes with history of pain and difficulty in overhead movements

Exclusion Criteria:

* Tumors of joint or bone.
* latex allergy
* Hypertension (i.e., resting systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg)
* Venous thrombotic disease
* Heart disease
* Respiratory disease;
* Dermatitis
* Psychiatric condition e.g depression,
* Recent history of shoulder fracture or humerus fracture.
* Rheumatoid arthritis.
* Osteoarthritis.
* Hyper-laxity of shoulder joint.
* Instability of shoulder
* Neuromuscular disorder
* Inflammatory disorder

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale | 2nd Week
  The 11-point numerical pain rating scale (NPRS) is a measure of pain in which patients rate their pain ranging from 0 (no pain) to 10 (worst imaginable pain), and it has been shown to have concurrent and predictive validity as a measure of pain intensity.
Shoulder pain and disability index | 2nd Week
  A shoulder pain and disability index (SPADI) is used to measure the pain and disability associated with shoulder pathology. The SPADI is a self-administered index consisting of 13 items divided into two subscales: pain and disability. The SPADI is responsive to change and accurately discriminates among patients who are improved or worsened.
Goniometer | 2nd Week
  A goniometer is an instrument that measures the available range of motion at a joint. The term Goniometry is derived from two Greek words, gonia, meaning "angle" and metron, meaning "measurement

CONTACTS AND LOCATIONS:
Overall Officials: Syed Shakil Ur Rehman, Principal Investigator — Riphah International University
Locations (1):
- Allied hospital Faisalabad, Pakistan, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Care IP, Renee Yacoub C. REHABILITATION FOLLOWING BICEPS BRACHII AND SUPRASPINATUS TENDINOPATHIES IN A 5-YEAR-OLD HAVANESE. 2019.
- [Background] Driller MW, Overmayer RG. The effects of tissue flossing on ankle range of motion and jump performance. Phys Ther Sport. 2017 May;25:20-24. doi: 10.1016/j.ptsp.2016.12.004. Epub 2016 Dec 12. PMID 28254581
- [Background] Cheatham SW, Baker R. Quantification of the Rockfloss(R) Floss Band Stretch Force at Different Elongation Lengths. J Sport Rehabil. 2020 Mar 1;29(3):377-380. doi: 10.1123/jsr.2019-0034. PMID 31094647
- [Background] 6. Kiefer BN, Lemarr KE, Enriquez CC, Tivener KA, Daniel T. A pilot study: perceptual effects of the voodoo floss band on glenohumeral flexibility. International Journal of Athletic Therapy and Training. 2017;22(4):29-33.
- [Background] Borda J, Selhorst M. The use of compression tack and flossing along with lacrosse ball massage to treat chronic Achilles tendinopathy in an adolescent athlete: a case report. J Man Manip Ther. 2017 Feb;25(1):57-61. doi: 10.1080/10669817.2016.1159403. Epub 2016 May 30. PMID 28855793
- [Background] Ekeberg OM, Bautz-Holter E, Keller A, Tveita EK, Juel NG, Brox JI. A questionnaire found disease-specific WORC index is not more responsive than SPADI and OSS in rotator cuff disease. J Clin Epidemiol. 2010 May;63(5):575-84. doi: 10.1016/j.jclinepi.2009.07.012. PMID 19836206
- [Background] Abbott JH, Schmitt J. Minimum important differences for the patient-specific functional scale, 4 region-specific outcome measures, and the numeric pain rating scale. J Orthop Sports Phys Ther. 2014 Aug;44(8):560-4. doi: 10.2519/jospt.2014.5248. Epub 2014 May 14. PMID 24828475
- [Background] 5. Parish E. Joint and Muscle Flossing.